CLINICAL TRIAL: NCT04170335
Title: Effects of Bariatric Surgery on Breast Density Improvement and Its Impact on Breast Cancer Risk in Morbidly Obese Patients
Brief Title: Effects of Bariatric Surgery on Breast Density Improvement and Impact on Breast Cancer Risk in Severe Obese Patients
Status: Withdrawn | Type: Observational
Why Stopped: No inclusion
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Raul Rosenthal, Chairman Department of Surgery, The Cleveland Clinic
Other Study IDs: FLA 18-057
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Morbid Obesity; Bariatric Surgery Candidate
Keywords: Breast cancer; Morbid obesity; Bariatric surgery; Mammography; Inflammatory markers
MeSH Terms: conditions — Breast Neoplasms; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric surgery group: Women older than age 40 and younger than age 74 undergoing primary bariatric surgery and having a BMI of ≥35 will be enrolled in this study. Pre operative and postoperative mammograms, inflammatory markers and breast cancer risk scores will be compared.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Patients selected and consented for elective bariatric surgery will undergo standard of care preoperative mammogram, as well as inflammatory markers measurements and breast cancer risk score calculation. Post bariatric surgery the patients will have follow up mammogram, inflammatory markers, and breast cancer risk score calculation

SUMMARY:
Breast cancer is the most common cancer in women in the US, and obese women have a 20% to 40% increase in the risk of developing breast cancer compared with normal-weight women. Bariatric surgery is now considered the first line option for weight loss management in morbidly obese patients with failure of medical treatment.

There is strong evidence that in early stages of cancer the breast undergoes inflammatory and subsequently density changes that are observable in mammography. The aforementioned alterations have been suggested to be magnified by obesity, potentially due to its pro-inflammatory state. The investigators hypothesized that rapid weight loss following bariatric surgery and henceforth the reduction of inflammatory stress in the breast tissue could potentially have a positive effect in improving breast density and consequently, reducing the risk of breast cancer. In this order of ideas, with this study, the investigators aim to evaluate how breast density is modified after bariatric surgery, and how it impacts the risk of developing breast cancer using The Breast Cancer Surveillance Consortium (BCSC) risk score and calculator in our population.

DETAILED DESCRIPTION:
This study is a prospective observational study involving patients selected for elective bariatric surgery. Thirty-five women older than age 40 and younger than age 74 undergoing primary bariatric surgery and having a BMI of ≥35 will be enrolled in this study. Patients with previous diagnosis of breast cancer, previous diagnosis of ductal carcinoma in situ (DCIS), previous breast augmentation and previous mastectomy will be excluded from the study. Patients selected and consented for elective bariatric surgery will be recruited in the Bariatric and Metabolic Institute at CCF, Weston FL and will undergo standard of care and additional measurements before and after surgery as explained below:

* A first mammogram study will be performed between two to four weeks before bariatric surgery, if the patient had a normal digital mammogram performed in the 12 months prior to bariatric surgery, it would be accepted as the first mammogram study. This mammogram is a part of the standard of care screening for this population group. Standard measurements will be assessed including the BI-RADS® breast density score (radiologic assessment of the density of breast tissue by a radiologist who interprets mammograms) and The LIBRA (Laboratory for Individualized Breast Radiodensity Assessment) software.
* A subsequent mammogram study (also part of the standard of care screening for this population group) will be performed one year after the date of the bariatric procedure, and standard measurements will be re-assessed, including re-stratification of BI-RADS and LIBRA.
* The mammogram results will be obtained through medical records. If a patient had done a mammogram at a non Cleveland Clinic facility, the investigator will ask them to sign an authorization form to allow Cleveland Clinic Florida to request for their mammography study from the previous year to the outside facility where it was done.
* Inflammatory markers including CRP, IGF1, IL6, TNF, will also be measured between two to four weeks before bariatric surgery as a part of the pre-surgical blood work up and, one year after the date of the bariatric procedure.

The inflammatory markers will be collected and processed as follows:

* CRP will be collected in a test tube containing lithium heparin (Green container). It will be delivered between two hours of collection to our institutional laboratory for processing.
* IGF1 will be collected in a test tube containing SST (Gold container). It will be delivered refrigerated between two hours of collection to our institutional laboratory for processing.
* IL6 will be collected in a test tube containing SST (Gold container). It will be delivered on ice ASAP upon collection to our institutional laboratory for processing.
* TNF will be collected in a test tube containing SST (Gold container). It will be delivered between two hours of collection to our institutional laboratory for processing.

  * Biometric measurements will be assessed before surgery and at the time of the subsequent mammogram (one year after surgery). It will include weight, height, BMI and Waist circumference.
  * Basic demographics and comorbidities (Diabetes Mellitus, Hypertension, pulmonary hypertension, sleep apnea, dyslipidemia, cardiovascular disease, chronic kidney disease, smoking status, alcohol use and hormonal replacement history) will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* women older than age 40 and younger than age 74 who qualify for bariatric surgery (BMI of ≥35 with at least one co-morbid condition), or BMI> 40

Exclusion Criteria:

* Patients with previous diagnosis of breast cancer, previous diagnosis of ductal carcinoma in situ (DCIS), previous breast augmentation and previous mastectomy will be excluded from the study

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women older than age 40 and younger than age 74 undergoing primary bariatric surgery selected and consented for elective bariatric surgery will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mammogram findings before and after intervention: BI-RADS | 12 months
  Mammogram findings according to the BI-RADS® breast density score (radiologic assessment of the density of breast tissue
Mammogram findings before and after intervention:LIBRA | 12 months
  Mammogram findings according to the The LIBRA (Laboratory for Individualized Breast Radiodensity Assessment) software
Inflammatory markers before and after intervention: C-reactive protein | 12 months
  Serum measurements of Inflammatory marker including C-reactive protein (CRP)
Inflammatory markers before and after intervention: Interleukin-6 | 12 months
  Serum measurements of Inflammatory marker including Interleukin-6 (IL-6)
Inflammatory markers before and after intervention: Insulin Growth Factor-1 (IGF-1) | 12 months
  Serum measurements of Inflammatory marker including Insulin Growth Factor-1 (IGF-1)
Inflammatory markers before and after intervention: Tumor Necrosis | 12 months
  Serum measurements of Inflammatory marker including Tumor Necrosis Factor (TNF)
Breast cancer risk calculation | 12 months
  Breast cancer risk calculation using The Breast Cancer Surveillance Consortium (BCSC) Risk Calculator
Biometric measurements: weight | 12 months
  Weight will be assessed before surgery and at one year after surgery.
Biometric measurements: Height | 12 months
  Height will be assessed before surgery and at one year after surgery.
Biometric measurements: Body mass index | 12 months
  Body mass index will be assessed before surgery and at one year after surgery.
Biometric measurements: Waist circumference. | 12 months
  Waist circumference. will be assessed before surgery and at one year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Raul Rosenthal, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steele CB, Thomas CC, Henley SJ, Massetti GM, Galuska DA, Agurs-Collins T, Puckett M, Richardson LC. Vital Signs: Trends in Incidence of Cancers Associated with Overweight and Obesity - United States, 2005-2014. MMWR Morb Mortal Wkly Rep. 2017 Oct 3;66(39):1052-1058. doi: 10.15585/mmwr.mm6639e1. PMID 28981482
- [Background] Vaysse C, Lomo J, Garred O, Fjeldheim F, Lofteroed T, Schlichting E, McTiernan A, Frydenberg H, Husoy A, Lundgren S, Fagerland MW, Richardsen E, Wist EA, Muller C, Thune I. Erratum: Inflammation of mammary adipose tissue occurs in overweight and obese patients exhibiting early-stage breast cancer. NPJ Breast Cancer. 2017 Sep 5;3:35. doi: 10.1038/s41523-017-0030-x. eCollection 2017. PMID 28884144
- [Background] Sun X, Glynn DJ, Hodson LJ, Huo C, Britt K, Thompson EW, Woolford L, Evdokiou A, Pollard JW, Robertson SA, Ingman WV. CCL2-driven inflammation increases mammary gland stromal density and cancer susceptibility in a transgenic mouse model. Breast Cancer Res. 2017 Jan 11;19(1):4. doi: 10.1186/s13058-016-0796-z. PMID 28077158
- [Background] McCormack VA, dos Santos Silva I. Breast density and parenchymal patterns as markers of breast cancer risk: a meta-analysis. Cancer Epidemiol Biomarkers Prev. 2006 Jun;15(6):1159-69. doi: 10.1158/1055-9965.EPI-06-0034. PMID 16775176
- [Background] Williams AD, So A, Synnestvedt M, Tewksbury CM, Kontos D, Hsiehm MK, Pantalone L, Conant EF, Schnall M, Dumon K, Williams N, Tchou J. Mammographic breast density decreases after bariatric surgery. Breast Cancer Res Treat. 2017 Oct;165(3):565-572. doi: 10.1007/s10549-017-4361-y. Epub 2017 Jun 28. PMID 28660430
- [Background] Keller BM, Chen J, Daye D, Conant EF, Kontos D. Preliminary evaluation of the publicly available Laboratory for Breast Radiodensity Assessment (LIBRA) software tool: comparison of fully automated area and volumetric density measures in a case-control study with digital mammography. Breast Cancer Res. 2015 Aug 25;17:117. doi: 10.1186/s13058-015-0626-8. PMID 26303303
- [Background] Schauer DP, Feigelson HS, Koebnick C, Caan B, Weinmann S, Leonard AC, Powers JD, Yenumula PR, Arterburn DE. Bariatric Surgery and the Risk of Cancer in a Large Multisite Cohort. Ann Surg. 2019 Jan;269(1):95-101. doi: 10.1097/SLA.0000000000002525. PMID 28938270